CLINICAL TRIAL: NCT06281886
Title: Induction Immuno-chemotherapy and Concurrent Chemoradiotherapy With or Without Apatinib in Unresectable, Locally Advanced Esophageal Squamous Cell Carcinoma: a Open-label, Randomized, Controlled Phase II Clinical Trial
Brief Title: Induction Immuno-chemotherapy and Concurrent Chemoradiotherapy With or Without Apatinib in Unresectable, Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10107
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma; Efficacy; Toxicity
Keywords: Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma; Induction immuno-chemotherapy; Concurrent chemoradiotherapy; Apatinib; Survival outcomes; Toxicity
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Radiotherapy; apatinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): Patients are planned to receive 2 cycles of induction immuno-chemotherapy plus apatinib, followed by concurrent chemoradiotherapy plus apatinib.
  Interventions: Drug: Induction Immunotherapy-Toripalimab; Drug: Induction Chemotherapy-Albumin-paclitaxel combined with cisplatin; Radiation: Radiotherapy; Drug: Apatinib; Drug: Capecitabine
- The control group (Active Comparator): Patients are planned to receive 2 cycles of induction immuno-chemotherapy, followed by concurrent chemoradiotherapy.
  Interventions: Drug: Induction Immunotherapy-Toripalimab; Drug: Induction Chemotherapy-Albumin-paclitaxel combined with cisplatin; Radiation: Radiotherapy; Drug: Capecitabine

INTERVENTIONS:
Drug: Induction Immunotherapy-Toripalimab — Toripalimab 240mg iv. drip, Q3W, 2 cycles
Drug: Induction Chemotherapy-Albumin-paclitaxel combined with cisplatin — Albumin-paclitaxel 260 mg/m2, administered on day 1, combined with cisplatin 25 mg/m2, administered on day 1,2,3.
Radiation: Radiotherapy — Thoracic radiotherapy at a total dose of 50Gy was delivered using the intensity modulated radiation therapy technique.
Drug: Apatinib — Oral apatinib 250mg once daily during induction therapy and concurrent chemoradiotherapy.
  Arms: The study group
Drug: Capecitabine — Oral capecitabine 1000 mg/m2, twice daily, on days 1-14, every 3 weeks, concurrently with radiotherapy
  Other Names: Chemotherapy concurrently with radiotherapy

SUMMARY:
This is an open-label, randomized, controlled phase II study evaluating induction immuno-chemotherapy and concurrent chemoradiotherapy with or without apatinib in unresectable, locally advanced esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
This is an open-label, randomized, controlled phase II study evaluating induction immuno-chemotherapy and concurrent chemoradiotherapy with or without apatinib in unresectable, locally advanced esophageal squamous cell carcinoma. In this study, patients are 1:1 randomized to either the study group or the control group. Patients in the study group will receive apatinib during induction immuno-chemotherapy and concurrent chemoradiotherapy. Patients in the control group will receive induction immuno-chemotherapy and concurrent chemoradiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with esophageal squamous cell carcinoma through pathological examination or cytological examination;
* Evaluated as locally advanced esophageal cancer that is unresectable through endoscopic ultrasound, imaging studies including barium swallow, CT scans of the neck, chest, and upper abdomen, MR imaging of the neck and chest, whole-body bone scan, or PET/CT, with staging ranging from T2-4, N0-3, M0-1 (M1 only includes patients with supraclavicular lymph node metastasis);
* Male or female aged between 18 and 80 years old;
* No prior chemotherapy, radiotherapy, surgery, targeted therapy, or immunotherapy;
* Expected survival of ≥12 weeks;
* ECOG performance status score of 0 or 1;
* Organ and bone marrow function meeting the following criteria: forced expiratory volume in 1 second (FEV1) ≥800 ml; absolute neutrophil count ≥1.5×109/L; platelet count ≥100×109/L; hemoglobin ≥90 g/L; serum creatinine clearance calculated according to the Cockcroft-Gault formula ≥50 mL/min (Cockcroft and Gault 1976); serum bilirubin ≤1.5 times the upper limit of normal (ULN); aspartate aminotransferase and alanine aminotransferase ≤2.5 times ULN;
* Signed and dated informed consent form is required before any study procedures are performed.

Exclusion Criteria:

* Participating in another clinical study concurrently, unless it is an observational (non-interventional) clinical study;
* Prior use of any targeted therapy or immunotherapy;
* Underwent major surgery (excluding vascular access) within 4 weeks before entering the study;
* Uncontrolled complications, including but not limited to persistent or active infections, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, arrhythmias, active peptic ulcer disease or gastritis, intestinal perforation, intestinal obstruction, active bleeding disorders, or psychiatric illness/social situations that would limit compliance with study requirements or impair the ability to provide written informed consent;
* Performance status score of 2-4;
* Any of the following organ and bone marrow dysfunctions: forced expiratory volume in 1 second (FEV1) <1000ml; absolute neutrophil count <1.5×109/L; platelet count <100×109/L; hemoglobin <90 g/L; serum creatinine clearance calculated according to the Cockcroft-Gault formula <50 mL/min (Cockcroft and Gault 1976); serum bilirubin >1.5 times the upper limit of normal (ULN); aspartate aminotransferase and alanine aminotransferase >2.5 times ULN;
* Conditions that may interfere with the assessment of the efficacy or safety of apatinib;
* Use of immunosuppressive drugs within 28 days before the first infusion of trastuzumab, excluding physiologic doses of inhaled corticosteroids; or systemic corticosteroids ≤10 mg/d of prednisone or equivalent;
* History of autoimmune diseases within the past 2 years;
* History of active or inflammatory bowel disease (such as Crohn's disease, ulcerative colitis);
* History of organ transplantation requiring immunosuppressive therapy;
* Receipt of attenuated live vaccines within 30 days before the study initiation or within 30 days after receiving trastuzumab;
* History of another primary malignancy within 5 years before starting trastuzumab, except adequately treated basal or squamous cell skin cancer or in situ cervical cancer;
* Pregnant or lactating females; or sexually active males or females of reproductive potential not using effective contraception methods.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate | 1 year
  From the first day of treatment to the day of progression or the day of death.

SECONDARY OUTCOMES:
Overall survival | 1 year
  It was calculated from the first day of treatment to the day of death.
Objective response rate | 1 year
  The proportion of patients evaluated as CR or PR
Local-regional progression-free survival | 1 year
  Local-regional progression-free survival refers to the period from the initiation of treatment until the occurrence of progression in the primary site or locoregional lymph node regions.
Incidence of Treatment-related Adverse Events | 1 year
  Adverse effects are graded according to the CTCAE 5.0 version, including multiple organs and tissues, such as gastrointestinal disease and symptom, cardiovascular disease, respiratory diseases and so on.
Score of Quality of Life Questionnare-Core 30 (The European Organization for Reasearch and Treatment of Cancer) | 1 year
  The evaluation of life quality
Distant metastasis-free survival | 1 year
  Distant metastasis-free survival refers to the period from the initiation of treatment until the appearance of metastasis in distant organs or tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Xu Y, Dong B, Zhu W, Li J, Huang R, Sun Z, Yang X, Liu L, He H, Liao Z, Guan N, Kong Y, Wang W, Chen J, He H, Qiu G, Zeng M, Pu J, Hu W, Bao Y, Liu Z, Ma J, Jiang H, Du X, Hu J, Zhuang T, Cai J, Huang J, Tao H, Liu Y, Liang X, Zhou J, Tao G, Zheng X, Chen M. A Phase III Multicenter Randomized Clinical Trial of 60 Gy versus 50 Gy Radiation Dose in Concurrent Chemoradiotherapy for Inoperable Esophageal Squamous Cell Carcinoma. Clin Cancer Res. 2022 May 2;28(9):1792-1799. doi: 10.1158/1078-0432.CCR-21-3843. PMID 35190815
- [Background] Conroy T, Galais MP, Raoul JL, Bouche O, Gourgou-Bourgade S, Douillard JY, Etienne PL, Boige V, Martel-Lafay I, Michel P, Llacer-Moscardo C, Francois E, Crehange G, Abdelghani MB, Juzyna B, Bedenne L, Adenis A; Federation Francophone de Cancerologie Digestive and UNICANCER-GI Group. Definitive chemoradiotherapy with FOLFOX versus fluorouracil and cisplatin in patients with oesophageal cancer (PRODIGE5/ACCORD17): final results of a randomised, phase 2/3 trial. Lancet Oncol. 2014 Mar;15(3):305-14. doi: 10.1016/S1470-2045(14)70028-2. Epub 2014 Feb 18. PMID 24556041
- [Background] Hulshof MCCM, Geijsen ED, Rozema T, Oppedijk V, Buijsen J, Neelis KJ, Nuyttens JJME, van der Sangen MJC, Jeene PM, Reinders JG, van Berge Henegouwen MI, Thano A, van Hooft JE, van Laarhoven HWM, van der Gaast A. Randomized Study on Dose Escalation in Definitive Chemoradiation for Patients With Locally Advanced Esophageal Cancer (ARTDECO Study). J Clin Oncol. 2021 Sep 1;39(25):2816-2824. doi: 10.1200/JCO.20.03697. Epub 2021 Jun 8. PMID 34101496
- [Background] Suntharalingam M, Winter K, Ilson D, Dicker AP, Kachnic L, Konski A, Chakravarthy AB, Anker CJ, Thakrar H, Horiba N, Dubey A, Greenberger JS, Raben A, Giguere J, Roof K, Videtic G, Pollock J, Safran H, Crane CH. Effect of the Addition of Cetuximab to Paclitaxel, Cisplatin, and Radiation Therapy for Patients With Esophageal Cancer: The NRG Oncology RTOG 0436 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2017 Nov 1;3(11):1520-1528. doi: 10.1001/jamaoncol.2017.1598. PMID 28687830
- [Background] Shinoda M, Ando N, Kato K, Ishikura S, Kato H, Tsubosa Y, Minashi K, Okabe H, Kimura Y, Kawano T, Kosugi S, Toh Y, Nakamura K, Fukuda H; Japan Clinical Oncology Group. Randomized study of low-dose versus standard-dose chemoradiotherapy for unresectable esophageal squamous cell carcinoma (JCOG0303). Cancer Sci. 2015 Apr;106(4):407-12. doi: 10.1111/cas.12622. Epub 2015 Mar 9. PMID 25640628
- [Background] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Background] Wang J, Yu JP, Wang JL, Ni XC, Sun ZQ, Sun W, Nie B, Jiang JT, Sun SP, Wu CP. [Pathologic response and changes of serum VEGF during chemoradiotherapy may predict prognosis in non-surgical patients with esophageal carcinoma]. Zhonghua Zhong Liu Za Zhi. 2016 Aug;38(8):589-95. doi: 10.3760/cma.j.issn.0253-3766.2016.08.005. Chinese. PMID 27531478
- [Background] Chu L, Chen Y, Liu Q, Liang F, Wang S, Liu Q, Yu H, Wu X, Zhang J, Deng J, Ai D, Zhu Z, Nie Y, Zhao K. A Phase II Study of Apatinib in Patients with Chemotherapy-Refractory Esophageal Squamous Cell Carcinoma (ESO-Shanghai 11). Oncologist. 2021 Jun;26(6):e925-e935. doi: 10.1002/onco.13668. Epub 2021 Feb 1. PMID 33393167
- [Background] Meng X, Wu T, Hong Y, Fan Q, Ren Z, Guo Y, Yang X, Shi P, Yang J, Yin X, Luo Z, Xia J, Zhou Y, Xu M, Liu E, Jiang G, Li S, Zhao F, Ma C, Ma C, Hou Z, Li J, Wang J, Wang F. Camrelizumab plus apatinib as second-line treatment for advanced oesophageal squamous cell carcinoma (CAP 02): a single-arm, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2022 Mar;7(3):245-253. doi: 10.1016/S2468-1253(21)00378-2. Epub 2022 Jan 6. PMID 34998471
- [Background] Chi D, Chen B, Guo S, Bai K, Ma H, Hu Y, Li Q, Zhu Y. Oral maintenance therapy using apatinib combined with S-1/capecitabine for esophageal squamous cell carcinoma with residual disease after definitive chemoradiotherapy. Aging (Albany NY). 2021 Mar 10;13(6):8408-8420. doi: 10.18632/aging.202652. Epub 2021 Mar 10. PMID 33713398
- [Background] Hu L, Sun F, Sun Z, Ni X, Wang J, Wang J, Zhou M, Feng Y, Kong Z, Hua Q, Yu J. Apatinib enhances the radiosensitivity of the esophageal cancer cell line KYSE-150 by inducing apoptosis and cell cycle redistribution. Oncol Lett. 2019 Feb;17(2):1609-1616. doi: 10.3892/ol.2018.9803. Epub 2018 Dec 6. PMID 30675220
- [Background] Hu L, Kong Z, Meng Q, Wang J, Zhou M, Yu J, Jiang X. The Safety and Efficacy of Apatinib Treatment in Addition to Concurrent Chemoradiotherapy in Patients with Nonoperative Locally Advanced Esophageal Squamous Cell Carcinoma. Med Sci Monit. 2020 Nov 27;26:e927221. doi: 10.12659/MSM.927221. PMID 33243967